CLINICAL TRIAL: NCT03517488
Title: A Phase 1 Multiple Dose Study to Evaluate the Safety and Tolerability of XmAb®20717 in Subjects With Selected Advanced Solid Tumors
Brief Title: A Study of XmAb®20717 in Subjects With Selected Advanced Solid Tumors
Acronym: DUET-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XmAb20717-01; DUET-2 (Other: Xencor, Inc.)
Record Dates: First submitted 2018-04-23; First posted 2018-05-07 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Melanoma; Breast Carcinoma; Hepatocellular Carcinoma; Urothelial Carcinoma; Squamous Cell Carcinoma of the Head and Neck; Renal Cell Carcinoma; Colorectal Carcinoma; Non-small Cell Lung Carcinoma; Gastric or Gastroesophageal Junction Adenocarcinoma; Endometrial Carcinoma; Mesothelioma; Neuroendocrine Carcinoma; Cervical Cancer; Small Cell Lung Carcinoma; Squamous Cell Carcinoma of the Anus; Castration-Resistant Prostate Carcinoma; Nasopharyngeal Carcinoma; Cholangiocarcinoma; Basal Cell Carcinoma; Ovarian Carcinoma; Fallopian Tube Carcinoma; Thymoma; Thymic Carcinoma; Squamous Cell Carcinoma of the Penis; Vulvar Carcinoma; Solid Tumors With Published Evidence of Anti-tumor Activity With Anti-PD1/PDL1 and/or Anti-CTLA4-directed Therapy; Malignant Adnexal Neoplasms; Non-squamous Cell Salivary Gland Carcinoma
Keywords: DUET-2; Melanoma; Triple Negative Breast Cancer; Hepatocellular Cancer; Urothelial Cancer; Renal Cell Cancer; Head and Neck Cancer; MSI-high Colorectal Cancer; MSI-high Endometrial Cancer; Non-small Cell Lung Cancer; Gastric Cancer; Gastroesophageal Junction Cancer; Mesothelioma; High-grade Neuroendocrine Cancer; Cervical Cancer; Small Cell Lung Cancer; Anal Cancer; Prostate Cancer; Nasopharyngeal Cancer; Bile Duct Cancer; Basal Cell Skin Cancer; Ovarian Cancer; Fallopian Tube Cancer; Malignant Adnexal Tumor; Thymus Cancer; Penile Cancer; Vulvar Cancer; Salivary Gland Cancer
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Transitional Cell; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Endometrial Neoplasms; Mesothelioma; Carcinoma, Neuroendocrine; Uterine Cervical Neoplasms; Small Cell Lung Carcinoma; Anus Neoplasms; Nasopharyngeal Carcinoma; Cholangiocarcinoma; Carcinoma, Basal Cell; Ovarian Neoplasms; Fallopian Tube Neoplasms; Thymoma; Vulvar Neoplasms; Triple Negative Breast Neoplasms; Liver Neoplasms; Head and Neck Neoplasms; Stomach Neoplasms; Prostatic Neoplasms; Nasopharyngeal Neoplasms; Bile Duct Neoplasms; Thymus Neoplasms; Penile Neoplasms; Salivary Gland Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XmAb20717 (Experimental): XmAb20717 administered by intravenous dosing on Days 1 and 15 of each 28-day cycle for a total of two cycles
  Interventions: Biological: XmAb20717

INTERVENTIONS:
Biological: XmAb20717 — Monoclonal bispecific antibody

SUMMARY:
This is a Phase 1, multiple dose, ascending dose escalation study to define a MTD/RD and regimen of XmAb20717, to describe safety and tolerability, to assess PK and immunogenicity, and to preliminarily assess anti-tumor activity of XmAb20717 in subjects with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of one of the following advanced solid tumors:

PART A (Dose Escalation Cohorts)

1. Melanoma;
2. Breast carcinoma that is estrogen receptor, progesterone receptor, and Her2 negative (triple-negative breast cancer; TNBC);
3. Hepatocellular carcinoma;
4. Urothelial carcinoma;
5. Squamous cell carcinoma of the head and neck;
6. Renal cell carcinoma (clear cell predominant type);
7. Microsatellite instability-high or mismatch repair deficient colorectal carcinoma or endometrial carcinoma;
8. Non-small cell lung carcinoma;
9. Gastric or gastroesophageal junction adenocarcinoma
10. Mesothelioma;
11. High-grade neuroendocrine carcinoma, including small cell carcinoma of the lung
12. Cervical cancer;
13. Squamous cell carcinoma of the anus

PART B (Dose Expansion Cohorts):

1. Melanoma
2. Renal cell carcinoma (clear cell predominant type)
3. Non-small cell lung carcinoma
4. Castrate-resistant adenocarcinoma of the prostate, defined as progressive disease after surgical castration, or progression in the setting of medical androgen ablation with a castrate level of testosterone (< 50 ng/dL)
5. Nasopharyngeal carcinoma
6. Cholangiocarcinoma
7. Basal cell carcinoma
8. Squamous cell carcinoma of the anus
9. Mesothelioma
10. Ovarian or fallopian tube carcinoma
11. Malignant adnexal neoplasms (including, but not limited to, sebaceous carcinoma, trichilemmal carcinoma, pilomatrix carcinoma, eccrine carcinoma, hidradenocarcinoma, adnexal carcinoma with divergent differentiation, papillary digital eccrine adenocarcinoma, microcystic adnexal carcinoma, and clear cell eccrine carcinoma)
12. Thymoma
13. Thymic carcinoma
14. Squamous cell carcinoma of the penis
15. Neuroendocrine carcinoma
16. Vulvar cancer
17. Non-squamous cell salivary gland carcinoma (except adenoid cystic carcinoma)
18. Subjects with other solid tumors for which there is published evidence of anti-tumor activity with anti-PD1/PDL1 and/or anti-CTLA4-directed therapy but for which there is no FDA-approved anti-PD1/PDL1 or CTLA4-directed checkpoint inhibitor treatment may be eligible for Part B after approval by the Medical Monitor.

    * All subjects' cancer must have progressed after treatment with all standard therapies or have no appropriate available therapies.
    * Subjects, except those with adenocarcinoma of the prostate, must have measurable disease by RECIST 1.1.
    * Have available adequate archival formalin-fixed paraffin-embedded block(s)/slides containing tumor or adequate pre-dose fresh tumor biopsy tissue
    * ECOG performance status of 0 - 1
    * Subjects with adenocarcinoma of the prostate must have evaluable disease (measurable or nonmeasurable lesions) by PCWG3.

Exclusion Criteria:

* Subjects currently receiving other anticancer therapies, with the exception of subjects with adenocarcinoma of the prostate, who may continue luteinizing hormone-releasing hormone (LHRH) analogue therapy.
* Treatment with any CTLA4 antibody within 6 weeks of the start of study drug.
* Treatment with nivolumab or any PDL1 or PDL2-directed antibody within 4 weeks of the start of study drug.
* Treatment with pembrolizumab within 4 - 12 weeks of the start of study drug (cohort dependent).
* Treatment with any other anticancer therapy within 2 weeks of the start of study drug (i.e., other immunotherapy, chemotherapy, radiation therapy, etc.). Subjects with prostate cancer may continue LHRH analogue therapy.
* A life-threatening (Grade 4) immune-mediated AE related to prior immunotherapy.
* Failure to recover from any immune-related toxicity from prior cancer therapy to ≤ Grade 1, except if previous immune-related endocrinopathy is medically managed with hormone replacement therapy only.
* Failure to recover from any other toxicity (other than immune-related toxicity) related to previous anticancer treatment to ≤ Grade 2.
* Have known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, ie, are without evidence of progression for at least 4 weeks by repeat imaging, are clinically stable, and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Active known or suspected autoimmune disease (except that subjects are permitted to enroll if they have vitiligo; type 1 diabetes mellitus or residual hypothyroidism due to an autoimmune condition that is treatable with hormone replacement therapy only; psoriasis, atopic dermatitis, or another autoimmune skin condition that is managed without systemic therapy; or arthritis that is managed without systemic therapy beyond oral acetaminophen and non-steroidal anti-inflammatory drugs).
* Has any condition requiring systemic treatment with corticosteroids, prednisone equivalents, or other immunosuppressive medications within 14 days prior to first dose of study drug (except that inhaled or topical corticosteroids or brief courses of corticosteroids given for prophylaxis of contrast dye allergic response are permitted).
* Receipt of an organ allograft.
* Prior treatment with any checkpoint inhibitor therapy regimen that targets both PD1/L1 and CTLA-4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability profile of XmAb20717 | 56 Days
  Treatment-related adverse events as assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Zequn Tang, MD, Study Director — Xencor, Inc.
Locations (17):
- United States (17):
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - UCLA Hematology-Oncology Clinic (Westwood), Los Angeles, California
  - University of California San Diego Moores Cancer Center, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Emory University, Atlanta, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - Karmanos Cancer Institute, Detroit, Michigan
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No